CLINICAL TRIAL: NCT05818423
Title: Brain Health Together: A Live-Streaming Group-Based Digital Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R44AG074727 (NIH); R44AG074727 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-04-18 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment; Cognitive Decline; Cognitive Deterioration; Cognitive Deficits, Mild; Cognitive Impairment, Mild
Keywords: Memory; Cognitive
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brain Health Academy (Experimental): Participant in this arm will watch expert videos on a wide range of brain health topics and will complete quizzes for 2.5 hours a week for 12 weeks (30 hours total)
  Interventions: Behavioral: Brain Health Academy
- Brain Health Together (Experimental): Participants in this arm will participate in online, live-streaming Moving Together classes (1 hour a week) and group brain health classes (1 hour a week) and will work 1-on-1 with a brain health coach to set personalized risk reduction goals (0.5 hours a week) for 12 weeks (30 hours total)
  Interventions: Behavioral: Brain Health Together
- Maintain Brain Health Together (Experimental): Participants in this arm will participate in the full Brain Health Together program for 12 weeks (30 hours) followed by weekly group classes and six 1-on-1 coaching sessions for another 12 weeks (additional 15 hours; 45 hours total)
  Interventions: Behavioral: Maintain Brain Health Together

INTERVENTIONS:
Behavioral: Brain Health Academy — The Brain Health Academy group will review online content about brain health (1 hour, 2 days/week for 12 weeks) and will complete a brief survey after each module to assess compliance (30 hours total).
  Arms: Brain Health Academy
Behavioral: Brain Health Together — The Brain Health Together group will participate in online, live-streaming, group-based Moving Together classes (1 hour/week); Brain Health education group classes (1 hour/week) and individual brain health coaching sessions (0.5 hours/week) for 12 weeks (30 hours total).
  Arms: Brain Health Together
Behavioral: Maintain Brain Health Together — The Maintaining Brain Health Together group will participate in the full Brain Health Together program (30 hours) for 12 weeks followed by weekly group classes and six individual coaching for an additional 12 weeks (additional 15 hours).
  Arms: Maintain Brain Health Together

SUMMARY:
The purpose of this study is to develop and test a comprehensive Brain Health Together program for older adults living with cognitive decline.

DETAILED DESCRIPTION:
Older adults with cognitive decline (including either mild cognitive impairment [MCI] or subjective cognitive decline [SCD]) represent a large market with important unmet needs. Approximately one in three older adults (18 million Americans) are currently living with cognitive decline, which places them at increased risk of developing Alzheimer's disease and related dementias (ADRD). There are no medications that can prevent development of dementia in people with cognitive decline; however, there is growing evidence that behavioral interventions targeting modifiable dementia risk factors-such as increasing physical activity and reducing social isolation-may help improve cognitive function and could potentially delay dementia onset. Preliminary results suggest that Moving TogetherTM program is associated with significant improvements in cognitive function, physical function, social isolation, and self-regulation as well as increased default mode network connectivity on pre/post resting state functional magnetic resonance imaging scans in people with cognitive decline. The investigators believe that these benefits would be even greater if Moving Together were combined with a comprehensive brain health coaching program.

ELIGIBILITY:
Inclusion Criteria:

* English language fluency;*
* live in U.S.;
* cognitive decline (subjective cognitive decline OR diagnosis of mild cognitive impairment in the past 12 months)
* ready to make lifestyle changes to improve brain health;
* have 2 or more brain health risk factors (e.g., low physical activity, depression, hypertension, diabetes, etc)
* have a desktop or laptop computer or iPad/tablet with a video camera;
* have broadband internet access;
* able to participate in online, live-streaming classes with two-way video

Exclusion Criteria:

Candidates meeting any of the exclusion criteria will not be eligible to participate.

Alzheimer's disease or dementia

- Major neurological disorder (e.g., Parkinson's disease, Multiple Sclerosis, amyotrophic Lateral Sclerosis)

* Schizophrenia or other psychotic disorder
* Autism or autism spectrum disorder
* Major mood or anxiety disorder that is not well-controlled (e.g., symptoms of depression or anxiety that made it hard to do daily tasks in past 6 months)
* Fracture of spine ("compression fracture") in the past 12 months
* Vertigo or severe dizziness in the past 12 months
* Severe vision or hearing impairment (e.g., unable to see and hear well enough to watch a movie on TV);
* Stroke or heart attack in the past 12 months
* Physical limitation that would restrict ability to participate (e.g., use wheelchair or walker to get around home, unable to stand up from sitting without assistance)
* Currently in another research study that could confound results of this study (e.g., drug study or other study to improve brain health)
* Previous participation in Moving Together or Brain Health Together
* Limited life expectancy (e.g., enrolled in hospice, undergoing cancer treatment)

If participants are not sure about certain conditions, they will be asked to describe their condition, and the research team will determine whether they meet eligibility criteria or not.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Maintain Your Brain Online Cognitive Test Battery-Change | Baseline and 3 months
  These are standard cognitive tests in three domains: attention, executive function, and learning/memory. individual test scores will be converted to standard scores using the means and standard deviations (SDs) of the study population. Tests within each domain will be averaged to create domain scores, and the three domain scores will then be averaged to create a single global composite score. Cognitive scores are standardized, mean=0, SD=1, expected range: -6 to +6 , highest score reflects the better outcome.
Alzheimer's Disease Risk Index - Short Form-Change (ANU-ADRI-SF) | Baseline and 3 months
  This is a validated measure that combines validated component measures of individual dementia risk factors and also provides a summary dementia risk score. It includes items related to demographics (age, sex, education), obesity, diabetes, hypercholesterolemia, head injury, depression, physical activity, cognitive activity, social isolation, alcohol consumption, smoking, pesticide exposure, and fish intake. Test scores with be combines to create a single global composite score. Cognitive scores are standardized, mean=0, SD=1, expected range: -6 to +6 , highest score reflects the better outcome.

SECONDARY OUTCOMES:
Physical activity-Change | Baseline and 3 months
  ANU-ADRI-SF assesses physical activity using the using the validated International Physical Activity Questionnaire short form. Participants are asked about time spent (days/week, minutes/day) doing vigorous physical activity, moderate physical activity, walking and sitting in the past 7 days, and responses are converted into metabolic equivalents per week. ANU-ADRI-SF - change range = -94 to +94, lower scores reflect the best outcome.
Depression-Change | Baseline and 3 months
  ANU-ADRI-SF assesses depressive symptoms using the validated 10-item version of the Center for Epidemiologic Studies-Depression Scale (CES-D). Participants are asked about feelings in the past week with response categories of 0 (<1/day), 1 (1-2 days), 2 (3-4 days) or 3 (5-7 days). Scores may range from 0 to 30, with higher scores indicating more depressive symptoms. NU-ADRI-SF - change range = -94 to +94, lower scores reflect the best outcome.
Loneliness / social isolation-Change | Baseline and 3 months
  The investigators will measure loneliness / social isolation using the validated measure 3-item UCLA Loneliness Scale, which consists of 3 items (lack companionship, feel left out, feel isolated) that are rated as 1 (hardly ever), 2 (some of the time), or 3 (often). Scores may range from 3 to 9, with higher scores reflecting greater loneliness.
Emotional well-being-Change | Baseline and 3 months
  Neuro-QOL v1.0 Positive Affect and Well-Being Short Form, which includes 9 items (e.g. sense of well-being, feeling hopeful, life was satisfying, etc.) with 5-point responses from never (1) to always (5). Scores may range from 9 to 45, with higher scores reflecting greater feelings of well-being.
Mind-body awareness-Change | Baseline and 3 months
  The investigators will measure mind-body awareness using the self-regulation sub-scale of the validated Multidimensional Assessment of Interoceptive Awareness version 2 (MAIA-2). The self-regulation sub-scale includes 4 items rated on a six-point Likert scale (0/never to 5/always) about the ability to regulate distress by paying attention to bodily sensations (e.g., "When I feel overwhelmed I can find a calm place inside.") Scores reflect the mean of responses (range 0 to 5), with higher scores indicating greater self-regulation.
Diet-Change | Baseline and 3 months
  The investigators will measure diet using the validated MIND diet score. The MIND diet is a hybrid of the Mediterranean and DASH (Dietary Approaches to Stop Hypertension) diets. It has 15 dietary components including 10 brain healthy foods (e.g., green leafy vegetables, berries) and 5 less healthy foods (e.g., red meat, fried/fast foods). The frequency of consumption for each item is scored as 0, 0.5 or 1, and the total MIND diet score is calculated by summing over the 15 components. Scores may range from 0 to 15, with higher scores reflecting better adherence to the MIND diet.
Obesity/weight-Change | Baseline and 3 months
  ANU-ADRI-SF includes questions about self-reported height and weight, which will be used to calculate body mass index (BMI). NU-ADRI-SF - change range = -94 to +94, lower scores reflect the best outcome.
Sleep-Change | Baseline and 3 months
  PROMIS Sleep Disturbance Short Form 4-item measure. The Investigators will measure sleep disturbance using the validated PROMIS Sleep Disturbance Short Form 4-item measure which asks about sleep quality and disturbance in the past 7 days on a 5-point Likert scale. Scores may range from 4 to 20 which higher scores indicating more sleep disturbance. In addition, we will include a single item from the Pittsburgh Sleep Quality Index on hours of sleep per night in the past month.
Self-efficacy/Confidence-Change | Baseline and 3 months
  Self-Efficacy for Managing Chronic Disease 6-item scale to measure self-efficacy for engaging in activities to support brain health. Each item is rated on an 11-point Likert scale from 0 (not at all confident) to 10 (totally confident). The score is the mean of the 6 items with higher scores reflecting higher self-efficacy.
Cognitive activity-Change | Baseline and 3 months
  Cognitive Activity Questionnaire (CAQ). The investigators will measure engagement in cognitive stimulating activities using a validated measure such as the Cognitive Activity Questionnaire (CAQ). The CAQ includes 11 items that ask how often individuals engage in various cognitive activities such as reading or playing games on a 6-point Likert scale (once a month/never to every day).
Alcohol-Change | Baseline and 3 months
  The investigators will measure alcohol consumption using 2 items in the ANU-ADRI that ask about frequency and amount of alcohol consumption.
Smoking-Change | Baseline and 3 months
  The investigators will assess smoking with standard questions about tobacco use ever and during the past 7 days
Global quality of life-Change | Baseline and 3 months
  The investigators will measure global quality of life using the validated PROMIS Scale v1.2 - Global Health. This scale includes 10 items rated on a 5-point Likert scale from 1 (poor) to 5 (excellent) and includes questions about overall self-rated health, overall quality of life, physical health, mental health, social relationships, fatigue and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Barnes, PhD, Principal Investigator — Primary Investigator
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Sharing permissions will be configured to ensure files containing PHI can only be accessed by authorized individuals. Two-step verification will be used as an additional safeguard against unauthorized access. Permissions will be updated when personnel roles change and they no longer need access to PHI or when they leave the research team.